CLINICAL TRIAL: NCT05153044
Title: Severe Acute Respiratory Syndrome CoV 2 Seroprevalence Survey and Vaccination Coverage in the Sickle Cell Population in Ile-De-France
Brief Title: Severe Acute Respiratory Syndrome CoV 2 COVID-19 Survey and Vaccination Coverage in the Sickle Cell Population in Ile-De-France
Acronym: COVIDO-DREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP211232
Record Dates: First submitted 2021-10-28; First posted 2021-12-10 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-09

CONDITIONS: Sickle Cell Disease
Keywords: seroprevalence; SARS-CoV-2; sickle cell
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- sickle cell children group (Other): sickle cell children group
  Interventions: Other: severe acute respiratory syndrome CoV-2 serology
- sickle cell adult group (Other): sickle cell adult group
  Interventions: Other: severe acute respiratory syndrome CoV-2 serology
- control children group (Other): control children group
  Interventions: Other: severe acute respiratory syndrome CoV-2 serology
- Vaccinated patients (No Intervention): Vaccinated patients

INTERVENTIONS:
Other: severe acute respiratory syndrome CoV-2 serology — diagnostic serology of severe acute respiratory syndrome-CoV-2 infection performed during the inclusion visit Regarding follow-up visits, only seropositive patients will be called for sampling, for serological follow-up at 3 months then 6 months.
  Arms: control children group; sickle cell adult group; sickle cell children group

SUMMARY:
The objective of this study is to determine the seroprevalence of severe acute respiratory syndrome-CoV-2 in unvaccinated sickle cell patients living in an area with high viral circulation and at risk of high viral transmission, after the 4th epidemic wave of COVID-19 in Ile-de -France, over a period of 3 months (for example, last quarter of 2021).

DETAILED DESCRIPTION:
Sickle cell disease is a very widespread genetic disease affecting 300,000 births worldwide, with a prevalence of one affected child for 1736 births in France, the most common genetic disease in France. France is the European country with the highest prevalence of the disease while Ile-de-France is the region with the highest prevalence of sickle cell disease and COVID-19. The medical management of sickle cell patients raises many challenges related to the complexity of their disease and the comorbidities that may be associated with their conditions (arterial hypertension, pulmonary arterial hypertension, nephropathy and renal failure, cerebral vasculopathy).Our seroprevalence study will focus on the sickle cell population living in an area with high circulation of severe acute respiratory syndrome-CoV-2; it will start after the 4th epidemic wave of COVID-19 during the vaccination campaigns, in order to collect on the one hand seroprevalence data (proportion of unvaccinated seropositive sickle cell patients) and persistence of humoral immunity (quantitative) after infection in unvaccinated subjects and on the other hand, to assess the vaccination coverage in this specific population (adults and adolescents) as well as its impact (occurrence of vaccine failures).

ELIGIBILITY:
Inclusion Criteria:

* Patient group = children with sickle cell disease:
* Children over 12 months of age and under 18 at the time of inclusion.
* Children with a major sickle cell syndrome (SS, "C gene and one sickle hemoglobin (S) gene", Sβ+, Sβ°, SE) followed in one of the centers of competence or reference for rare diseases (CRMR) "Major Sickle Cell Syndromes, Thalassemias and Other Rare Pathologies of Red Blood Cell and Erythropoiesis "from Ile de France.
* Children not subject to legal protection measures.
* Children affiliated to a French social security scheme
* Informed consent signed by one of the two parents.

Group of adults with sickle cell disease:

* Patients over 18 years of age at the time of inclusion (male, female).
* Patients with a major sickle cell syndrome (SS, "C gene and one sickle hemoglobin (S) gene", Sβ+, Sβ°, SE) followed in one of the centers of competence or reference for rare diseases (CRMR) "Major Sickle Cell Syndromes, Thalassemias and Other Rare Pathologies of Red Blood Cell and Erythropoiesis "from Ile de France.
* Patients not subject to legal protection measures.
* Patients affiliated to a French social security scheme
* Informed consent signed

Child-control group:

* Children over 12 months old and under 18 years old at the time of inclusion.
* Children without sickle cell disease
* Children monitored for asthma or with a history of asthma.
* Children not subject to legal protection measures.
* Children affiliated to a French social security scheme
* Informed consent signed by one of the two parents.

Exclusion Criteria:

* Patient group = sickle cell children :
* Infants under 12 months of age.
* Other haemoglobinopathies and heterozygous Haemoglobin AS or AC patients.
* Children already in a treatment protocol or in the exclusion period from a previous investigation.
* Children on state medical assistance

Adult sickle cell group :

* Other haemoglobinopathies and heterozygous AS or AC patients.
* Patients already on a treatment protocol or in the exclusion period from a previous investigation.
* Pregnant or lactating women.
* Patients on state medical assistance

Child control group :

* Infants under 12 months of age and adults over 18 years of age.
* Children already in a treatment protocol or in the exclusion period from a previous study.
* Children on state medical assistance

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-09-10 (Estimated)

PRIMARY OUTCOMES:
The positivity of total anti-SARS-CoV-2 blood Ig will be determined by the presence of anti-spike protein Ig G and / or anti-nucleocapsid Ig G (post-infectious COVID-19 humoral immunity). | 9 months
  To determine the seroprevalence of SARS-CoV-2 after the 4th epidemic wave in unvaccinated sickle cell patients (children and adults), living in an area with high viral circulation of SARS-CoV-2 and high risk of viral transmission, in Ile-De-France.

SECONDARY OUTCOMES:
The positivity anti-SARS-CoV-2 serology and anti-spike antibody titre from M0 to M6. | 9 months
  Compare the seroprevalence and decrease in antibodies (initial M0 titre and duration of persistence at M3-M6) in unvaccinated patients with a history of COVID-19 infection between the group of children with sickle cell disease, the group of children non-sickle cell control patients and the group of adults with sickle cell disease.
Negativity of anti-SARS-CoV-2 serology at M3 and M6. | 3 and 6 months
  Investigation of factors associated with a faster loss of anti-SARS-CoV-2 blood antibodies (age, sex, genotype, splenectomy, transplants, treatment with hydroxyurea) in unvaccinated sickle cell patients with a history of COVID-19 infection.
COVID-19 infection (nasopharyngeal RT-PCR Reverse transcription-polymerase chain reaction positivity and/or COVID-19 anti-SARS-CoV-2 serology). | 9 months
  Assessing factors associated with the risk of COVID-19 infection (epidemiological, environmental and sickle cell disease related) in sickle cell patients.
Intensive care unit admission for COVID-19. | 9 months
  Assessing factors associated with a severe form of COVID-19 infection among sickle cell patients.
Proportion of patients vaccinated among the patients interviewed and included in the study. | 9 months
  Determine the vaccination coverage rate of the sickle cell population (according to age groups) over a period of 3 months, after the 4th epidemic wave of 2021.
Occurrence of post-vaccine side effects (fever, pain, vaso-occlusive crisis, myocarditis, others) | 9 months
  List the occurrence of declared side effects.
Proportion of COVID-19 infection occurring in vaccinated patients. | 9 months
  Determine the incidence rate of COVID-19 infection in vaccinated patients (vaccine failure rate)

REFERENCES:
- [Background] Menapace LA, Thein SL. COVID-19 and sickle cell disease. Haematologica. 2020 Nov 1;105(11):2501-2504. doi: 10.3324/haematol.2020.255398. No abstract available. PMID 33131239
- [Background] Vilela TS, Braga JAP, Loggetto SR. Hemoglobinopathy and pediatrics in the time of COVID-19. Hematol Transfus Cell Ther. 2021 Jan-Mar;43(1):87-100. doi: 10.1016/j.htct.2020.11.002. Epub 2020 Dec 2. PMID 33289008
- [Background] Wajnberg A, Amanat F, Firpo A, Altman DR, Bailey MJ, Mansour M, McMahon M, Meade P, Mendu DR, Muellers K, Stadlbauer D, Stone K, Strohmeier S, Simon V, Aberg J, Reich DL, Krammer F, Cordon-Cardo C. Robust neutralizing antibodies to SARS-CoV-2 infection persist for months. Science. 2020 Dec 4;370(6521):1227-1230. doi: 10.1126/science.abd7728. Epub 2020 Oct 28. PMID 33115920